CLINICAL TRIAL: NCT06934954
Title: Adapted Early Adolescent Skills for Emotions (EASE) to Decrease Psychological Distress Among Urban Youth and Caregivers in NYC: a Pilot Study
Brief Title: Early Adolescent Skills for Emotions
Acronym: EASE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The New School (Other)
Responsible Party: Principal Investigator, Adam Brown, Ph.D., Principal Investigator, The New School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EASE; 000001 (Other Grant/Funding Number: New York City Mayors Office Community Mental Health)
Record Dates: First submitted 2025-03-27; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Community Mental Health Services
Keywords: Youth Mental Health; Adolescent Mental Health; Community Mental Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EASE Intervention (Experimental): EASE targets psychological distress in adolescents ages 10 to 15 years old through seven group sessions with adolescents and three group sessions with the adolescents' caregivers. Each session is 90 minutes, and adolescents learn and engage in strategies that progress in complexity throughout the intervention. Through EASE, adolescents learn how to identify their emotions, distress-related physical arousal, slow breathing as a healthy coping strategy, behavioral activation to engage in meaningful activities, and problem-solving skills. RCTs have indicated the scalability and efficacy of EASE in LMICs like Lebanon and Syria. To prepare for pilot implementation, researchers from The New School Center for Global Mental Health collected feedback from community partners on EASE in 2024. Based on community recommendations, EASE was adapted for the current study.
  Interventions: Behavioral: EASE

INTERVENTIONS:
Behavioral: EASE — This is the first time EASE is being used in New York to support youth community mental health.

SUMMARY:
The EASE program is an existing, evidence-based program/intervention (originally developed by the WHO), and this study is limited to evaluating the local implementation of this program.

The aims of this pilot study are to:

* Assess the acceptability and feasibility of training and supervision of EASE Helpers (community staff members) through an adapted EASE training.
* Evaluate possible problems of recruitment, intervention delivery, and participant retention.
* Assess the feasibility of EASE being delivered via a partnership between researchers and community members.
* Evaluate implementation of EASE via the RE-AIM (Reach, Effectiveness, Adoption, Implementation, and Maintenance) framework

A mixed-methods design with qualitative and quantitative approaches will be used to assess these objectives.

DETAILED DESCRIPTION:
Despite the growing need for adolescent mental health services in the US, access to treatment has remained especially inequitable for ethnic minorities. Studies have identified socio-ecological barriers, such as stigma, caregiver attitudes, and income, that contribute to a number of disparities between ethnically minoritized adolescents and their white counterparts. Although there is support for evidence-based psychotherapies in improving youth mental health outcomes generally, the mental health burden and structural inequities faced by ethnically minoritized adolescents call for novel approaches that may address some of the challenges and bridge the services and treatment gap.

One approach that is becoming increasingly studied globally is task-sharing mental health interventions. Task-sharing often refers to brief and non-specialist-delivered versions of evidence-based psychological treatments for people with mildly to moderately severe mental health symptoms, especially in under resourced settings and low- and middle-income countries (LMICs). Randomized controlled trials (RCTs) have indicated that scalable mental health interventions are effective in reducing symptoms of distress and post-traumatic symptomatology across different populations and contexts at follow-up assessments.

Although there is now considerable work evaluating the potential benefits of task-sharing interventions globally, this approach is somewhat newer in the US. However, burgeoning work in the US is beginning to show the feasibility of such intervention with adults. The New School Center for Global Mental Health has also conducted adaptations, training, and program evaluations for task-sharing interventions like the World Health Organization's (WHO) Problem Management Plus (PM+) for adult community members in NYC since 2020. Initial evaluations have indicated the acceptability, feasibility, and utility of PM+ in the NYC context. Given the evidence-based support for task-sharing interventions for adults and the treatment and services gap for ethnically minoritized adolescents in NYC, the investigators would like to evaluate how well a WHO task-sharing intervention for adolescents - Early Adolescent Skills for Emotions (EASE) - works in community-based organizations in NYC.

EASE targets psychological distress in adolescents ages 10 to 15 years old through seven group sessions with adolescents and three group sessions with the adolescents' caregivers. Each session is 90 minutes, and adolescents learn and engage in strategies that progress in complexity throughout the intervention. Through EASE, adolescents learn how to identify their emotions, distress-related physical arousal, slow breathing as a healthy coping strategy, behavioral activation to engage in meaningful activities, and problem-solving skills. RCTs have indicated the scalability and efficacy of EASE in LMICs like Lebanon and Syria.

To prepare for pilot implementation, researchers from The New School Center for Global Mental Health collected feedback from community partners on EASE in 2024. Based on community recommendations, adaptations to EASE's manual activities/strategies and storybook were made to improve EASE's acceptability, relevance, and accessibility.

The proposed study aims to implement this culturally-adapted version of EASE to urban youth and caregivers in NYC in collaboration with CBOs identified by the NYC Mayor's Office of Community Mental Health (OCMH). Youth/adolescents in this study are defined as children ages 10 to 15 years old. Caregivers in this study are defined as the adults who regularly take care of adolescent(s) 10 to 15 years olds, typically in their home settings. All caregivers that are asked to provide consent for a child's participation in the study will also be the child's legally authorized representative (i.e., parent or legal guardian). The person providing permission for the child to participate in the study must confirm that they are the adolescent's parent or legal guardian. Decisions can be made for adolescents and children by their caregivers if the caregivers are also the adolescents' legally authorized representative. In doing so, the investigators hope to examine the effectiveness, feasibility, acceptability, and utility for implementing EASE in the US and collect additional feedback to improve the adaptation to better bridge the mental health services and treatment gap for urban youth.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents

  * 10-15 years old
  * English-speaking
  * Has obtained parental permission from a legally authorized representative (e.g. legal guardian).

    ○ Caregiver
  * English-speaking
  * Is a caretaker of a child ages 10-15 years old, meaning they regularly take care of a child
  * Adults who are above the age of 18 who meet the above criteria can participate.

Exclusion Criteria:

* The program is not intended for adolescents and caregivers who are experiencing severe cognitive impairments and/or have an imminent risk of suicide/acute protection needs.

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pediatric Symptom Checklist Youth Report (Y-PSC) | 8 months
  For youth participants: The Pediatric Symptom Checklist Youth Report (Y-PSC) is a 35 item questionnaire that helps identify and assess changes in emotional and behavioral problems in children. Participants are to respond to how often they have had certain thoughts, feelings, and experiences listed in the questionnaire in the past 2 weeks with the options "never", "sometimes", and "often".

SECONDARY OUTCOMES:
Patient Health Questionnaire - Adolescent Version (PHQ-A) | 8 months
  For youth participants: The PHQ-A assesses degree of depression severity for adolescents via questionnaire. Participants are to respond to how often they have had certain thoughts and feelings listed in the questionnaire in the past 2 weeks with the options "not at all", "several days", "more than half the days", and "nearly every day".
Warwick Edinburgh Well-being Scale (WEMWBS) | 8 months
  For youth participants: The WEMWBS is a 14-item scale of positively worded statements covering feeling and functioning aspects of mental wellbeing. Participants are to respond to how often they have had certain thoughts and feelings listed in the questionnaire in the past 2 weeks with the options "none of the time", "rarely", "some of the time", "often", and "all of the time".
Impairment of Daily Function | 8 months
  For youth participants: The Impairment of daily functioning tool evaluates an individual's ability to perform basic and instrumental activities of daily living. Participants are to respond to how difficult it is generally to complete some daily tasks with the options "no difficulty", "little difficulty", "moderate difficulty", "a lot difficulty", and "often can't do task".
Psychological Sense of School Membership (PSSM) | 8 months
  For youth participants: The Psychological Sense of School Membership is an 18-item tool that measure adolescent students' perceived belonging or psychological membership in the school environment. Participants are to respond to the statements in the questionnaire on a scale. The minimum value of the scale is 1 and the maximum value of the scale is 5. 1 refers to not at all true and 5 refers to completely true. Whether a higher score means a better or worse outcome depends on whether the questionnaire statement needs to be reverse-coded.
Parental Stress Scale (PSS) | 8 months
  For caregiver participants: The Parental Stress Scale (PSS) is an 18-item questionnaire assessing parents' feelings about their parenting role. Participants are to answer statements on a scale. The minimum value is 1 (strongly disagree) and the maximum value is 5 (strongly agree). Whether a higher score means a better or worse outcome depends on whether the questionnaire statement needs to be reverse-coded.
Alabama Parenting Questionnaire (APQ) | 8 months
  For caregiver participants: The Alabama Parenting Questionnaire (APQ) is a self-report assessment tool designed to measure five key dimensions of parenting that are related to child behavioral problems. Participants are to respond to how often statements of experiences described in the questionnaire typically occur in their home. The options are "never", "almost never", "sometimes", "often", and "always".
Patient Health Questionnaire (PHQ-9) | 8 months
  For caregiver participants: The PHQ-9 (Patient Health Questionnaire-9) is a self-report questionnaire used to assess the presence and severity of depressive symptoms. Participants are to respond to how often they have had certain thoughts and feelings listed in the questionnaire in the past 2 weeks with the options "not at all", "several days", "more than half the days", and "nearly every day".
Generalized Anxiety Disorder Assessment (GAD-7) | 8 months
  For caregiver participants: The Generalized Anxiety Disorder Assessment (GAD-7) is a seven-item instrument that is used to measure or assess the severity of generalised anxiety disorder (GAD). Participants are to respond to how often they have had certain thoughts and feelings listed in the questionnaire in the past 2 weeks with the options "not at all", "several days", "more than half the days", and "nearly every day".
Kessler's Psychological Distress Scale (K6+) | 8 months
  For caregiver participants: The Kessler Psychological Distress Scale (K6+) is a 6-item self-report measure of psychological distress intended to be used as a quick tool to assess risk for serious mental illness in the general population. Participants are to respond to how often they have had certain thoughts and feelings listed in the questionnaire in the past 30 days with the options "all of the time", "most of the time", "some of the time", "a little of the time", and "none of the time".

CONTACTS AND LOCATIONS:
Overall Officials: Adam Brown, PhD, Principal Investigator — The New School
Locations (1):
- The New School Center for Global Mental Health, New York, New York, United States

REFERENCES:
- [Background] Brown FL, Taha K, Steen F, Kane J, Gillman A, Aoun M, Malik A, Bryant R, Sijbrandij M, El Chammay R, Servili C, van Ommeren M, Akhtar A, Zoghbi E; EASE Intervention Development, Training Team; Jordans MJD; STRENGTHS Consortium. Feasibility randomised controlled trial of the Early Adolescent Skills for Emotions psychological intervention with young adolescents in Lebanon. BMC Psychiatry. 2023 Mar 1;23(1):131. doi: 10.1186/s12888-023-04571-9. PMID 36858980
- [Background] Castro-Ramirez F, Al-Suwaidi M, Garcia P, Rankin O, Ricard JR, Nock MK. Racism and Poverty are Barriers to the Treatment of Youth Mental Health Concerns. J Clin Child Adolesc Psychol. 2021 Jul-Aug;50(4):534-546. doi: 10.1080/15374416.2021.1941058. Epub 2021 Aug 2. PMID 34339320
- [Background] Fan Q, DuPont-Reyes MJ, Hossain MM, Chen LS, Lueck J, Ma P. Racial and ethnic differences in major depressive episode, severe role impairment, and mental health service utilization in U.S. adolescents. J Affect Disord. 2022 Jun 1;306:190-199. doi: 10.1016/j.jad.2022.03.015. Epub 2022 Mar 14. PMID 35301042
- [Background] Dawson KS, Watts S, Carswell K, Shehadeh MH, Jordans MJD, Bryant RA, Miller KE, Malik A, Brown FL, Servili C, van Ommeren M. Improving access to evidence-based interventions for young adolescents: Early Adolescent Skills for Emotions (EASE). World Psychiatry. 2019 Feb;18(1):105-107. doi: 10.1002/wps.20594. No abstract available. PMID 30600639
- [Background] Alegria M, Vallas M, Pumariega AJ. Racial and ethnic disparities in pediatric mental health. Child Adolesc Psychiatr Clin N Am. 2010 Oct;19(4):759-74. doi: 10.1016/j.chc.2010.07.001. PMID 21056345
- [Background] Weersing VR, Gonzalez A, Hatch B, Lynch FL. Promoting Racial/Ethnic Equity in Psychosocial Treatment Outcomes for Child and Adolescent Anxiety and Depression. Psychiatr Res Clin Pract. 2022 Sep 9;4(3):80-88. doi: 10.1176/appi.prcp.20210044. eCollection 2022 Fall. PMID 36177440
- [Background] Lu W, Todhunter-Reid A, Mitsdarffer ML, Munoz-Laboy M, Yoon AS, Xu L. Barriers and Facilitators for Mental Health Service Use Among Racial/Ethnic Minority Adolescents: A Systematic Review of Literature. Front Public Health. 2021 Mar 8;9:641605. doi: 10.3389/fpubh.2021.641605. eCollection 2021. PMID 33763401
- [Background] Jordans MJD, Brown FL, Kane J, Taha K, Steen F, Ali R, Elias J, Meksassi B, Aoun M, Greene CM, Malik A, Akhtar A, van Ommeren M, Sijbrandij M, Bryant R; STRENGTHS consortium. Evaluation of the Early Adolescent Skills for Emotions (EASE) intervention in Lebanon: A randomized controlled trial. Compr Psychiatry. 2023 Nov;127:152424. doi: 10.1016/j.comppsych.2023.152424. Epub 2023 Sep 16. PMID 37748283
- [Background] Bryant RA, Malik A, Aqel IS, Ghatasheh M, Habashneh R, Dawson KS, Watts S, Jordans MJD, Brown FL, van Ommeren M, Akhtar A. Effectiveness of a brief group behavioural intervention on psychological distress in young adolescent Syrian refugees: A randomised controlled trial. PLoS Med. 2022 Aug 12;19(8):e1004046. doi: 10.1371/journal.pmed.1004046. eCollection 2022 Aug. PMID 35960704

DOCUMENTS (1):
  • Informed Consent Form (2025-03-12): https://cdn.clinicaltrials.gov/large-docs/54/NCT06934954/ICF_000.pdf